CLINICAL TRIAL: NCT06588517
Title: A Randomized, Open-Label, Two-Period, Double-Crossover Comparative Study on the Pharmacokinetics of Pirfenidone Modified-Release Tablets and Pirfenidone Tablets in Healthy Chinese Subjects Under Fed Conditions
Brief Title: Comparative Pharmacokinetic(PK) Study of Pirfenidone Modified-Release Tablets and Pirfenidone Tablets in Healthy Subjects Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Overseas Pharmaceuticals, Ltd. (Industry)
Collaborators: Shanghai ShouYan Clinical Development Co.,Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: YY-BFNT-2024
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Pirfenidone; Modified-Release; Idiopathic pulmonary fibrosis; Healthy Volunteers
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group T (Experimental): take the tablet under fed condition ,1 tablet at a time, once a day.Test product (T): Pirfenidone Modified-
  Release Tablets Strength: 600 mg/tablet Batch No.:
  08532 Content: 600 mg/tablet Valid to: January/2025 Storage Conditions: sealed at normal temperature (10-30°C) Manufacturer: Overseas Pharmaceuticals, Ltd.
  Interventions: Drug: Pirfenidone Modified-Release Tablets
- Group R (Active Comparator): take the tablet under fed condition ,1 tablet at a time, three times a day.Reference product (R): Pirfenidone Tablets Strength: 200 mg/tablet Batch No.: 0239 Content: 200 mg/tablet Valid to: September 2026 Storage Conditions: sealed at room temperature Manufacturer: Shionogi & Co., Ltd..
  Interventions: Drug: Pirfenidone Tablets

INTERVENTIONS:
Drug: Pirfenidone Modified-Release Tablets — take the tablet under fed condition, 1 tablet at a time, once a day.
  Arms: Group T
Drug: Pirfenidone Tablets — ake the tablet under fed condition, 1 tablet at a time, three times a day.
  Arms: Group R

SUMMARY:
A Randomized, Open-Label, Two-Period, Double-Crossover Comparative Study on the Pharmacokinetics of Pirfenidone Modified-Release Tablets and Pirfenidone Tablets in Healthy Chinese Subjects under Fed Conditions Primary objective: To evaluate the bioequivalence of test product and reference product by comparing their plasma concentrations and main PK parameters by oral administration in healthy Chinese subjects under fed conditions using Pirfenidone Modified-Release Tablets (strength: 600 mg/tablet) developed by Overseas Pharmaceuticals, Ltd. as the test product and Pirfenidone Tablets (trade name: Pirespa®, strength: 200 mg/tablet) produced by Shionogi & Co., Ltd. as the reference product. Secondary objective: To evaluate the safety of Pirfenidone Modified-Release Tablets (test product) and Pirfenidone Tablets (reference product) after oral administration in healthy Chinese subjects under fed conditions.

DETAILED DESCRIPTION:
It is designed to be a single-center, randomized, open-label, two-period, double-crossover trial. All subjects must sign an informed consent form (ICF) prior to participation in the trial. Twenty-four (24) eligible healthy subjects (male and female, with an appropriate sex ratio) screened through physical examination from D-14 to D-1 of dosing will be randomized into Group T-R and Group R-T, with 12 subjects in each group. The enrolled subjects will be admitted to phase I ward of the clinical study site 1 day before medication in each period and fasted for more than 10 h before medication.

On the morning of medication, after the collection of blank blood samples within 60 minutes before administration, both group will have a standard breakfast that completed within 10 min±30 s. Group T will orally take 1 tablet of Pirfenidone Modified-Release Tablets (600 mg/tablet, Overseas Pharmaceuticals, Ltd.) developed by Overseas Pharmaceuticals, Ltd. in 12 minutes after starting a standard breakfast ; Group R will orally take 3 tablet of Pirfenidone Modified-Release Tablets (600 mg/tablet, Overseas Pharmaceuticals, Ltd.) under fed condition（The first tablet should be taken in 12 minutes after the start of a standard breakfast, the second tablet should be taken in 30 minutes (±30 s) after the start of a standard lunch, and the third tablet should be taken in 30 minutes (±30 s) after the start of a standard dinner）.

Standard lunch is served 4 h after administration, standard dinner 10 h later, water is prohibited before and within 1 h after administration (except 240 mL water for medication), and unified diet is required during the trial.

Unified diet is required during the trial. The trial method in period II is the same as that in period I, with a washout period of 6 days.

PK blood sampling and blood sample processing:

Cubital venous blood will be collected at 31 time points: before administration (0 h) and 0.25 h, 0.50 h, 1.00 h, 1.50 h, 2.00 h, 3.00 h, 4.00 h, 4.50 h, 5.00 h, 6.00 h, 7.00 h, 7.50 h, 8.00 h, 9.00 h, 10.00 h, 10.25 h, 10.50 h, 11.00 h, 11.50 h, 12.00 h, 12.50 h, 13.00 h, 14.00 h, 16.00 h, 18.00 h, 20.00 h, 24.00 h, 28.00 h, 36.00 h and 48.00 h after administration of each period.

Four milliliters (4 mL) (scale of 4 mL should be pre-marked on the blood collection tube) will be drawn and placed in a labeled EDTA-2K anticoagulant tube. The collection, processing and storage procedures of biological samples are subject to the final sample operation manual. Sitting vital signs (including respiratory rate, body temperature, pulse rate, and sitting blood pressure) will be measured within 1 h before administration and at 2 ± 0.5 h, 8 ± 0.5 h, 24 ± 0.5 h and 48 ± 1 h after administration. Subjects should receive physical examination, vital signs, ECG, and laboratory-related tests on D2 after the last dose. The subjective feelings of subjects as well as possible adverse reactions (ARs) and adverse events (AEs) occurred during the trial should be observed and inquired. All subjects will be followed up for 7 days after the end of the last dose to inquire the occurrence of any subsequent AEs. If occurred, AEs should be recorded and followed up. An AE emerged during the trial should be followed up until it is resolved.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects over the age of 18 years (including those aged 18 years), with an appropriate sex ratio;
2. Male subjects with a body weight ≥ 50.0 kg, and female subjects with a body weight ≥ 45.0 kg; BMI (BMI = body weight (kg)/[height (m)]2) within the range of 19-26.0 kg/m2 (including the critical value);
3. Subjects with good health conditions, no clinically significant medical history in respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, and mental system;
4. Subjects (including partners) who have no plans of pregnancy and voluntarily take appropriate contraceptive measures from the date of signing the informed consent (14 days before signing the informed consent for female subjects) to 6 months after the end of the study;
5. Subjects who are able to communicate well with the investigator and understand and adhere to the study requirements. Subjects who fully understand the objective, nature, method and possible ARs of the trial, voluntarily act as subjects, and sign the ICF before any study procedures are started;

Exclusion Criteria:

1. Patients with an allergic history to the study drug or its excipients (such as lactose), or an allergic history to drug, food , pollen or a specific allergic history (asthma, allergic rhinitis, eczema);
2. Patients with a history of photosensitivity and existing skin irritation symptoms such as rash and pruritus;
3. Subjects who have special dietary requirements and cannot accept a unified diet;
4. Subjects with a history of dysphagia or any gastrointestinal disorder affecting drug absorption;
5. Subjects who cannot tolerate venipuncture and have a history of fear of needles and hemophobia;
6. Subjects with clinically significant hematological, endocrine, cardiovascular, hepatic, renal and pulmonary disorders that may affect drug absorption, distribution, metabolism and excretion;
7. Subjects with a surgical history or taking the study drug or participating in other drug clinical trials within 3 months prior to the study;
8. Subjects with blood donation or massive blood loss (> 450 mL) within 3 months before the study;
9. Subjects taking special diet (including pitaya or grapefruit and products containing grapefruit ingredients) or having strenuous exercise within 7 days before taking the study drug, or having other factors affecting drug absorption, distribution, metabolism and excretion;
10. Subjects administered with any prescription drugs, over-the-counter, herbal, or health products within 14 days prior to taking the study drug;
11. Regular drinkers within 6 months prior to the study, i.e., drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirit containing 40% alcohol or 150 mL of wine);
12. Subjects smoking more than 5 cigarettes per day in the first 3 months of the study; Or positive results of tobacco test;
13. Subjects who have consumed chocolate, any caffeine-containing, or xanthine-rich food or beverage, such as coffee, strong tea, and cola 48 h before taking the study drug;
14. Subjects having taken any alcohol-containing products within 48 h before taking the study drug, or having a positive result for alcohol screening;
15. Female subjects with positive pregnancy
16. Subjects positive for HBsAg, HCV-Ab, anti-HIV or primary syphilis screening;
17. Subjects positive for drug screening or with a history of drug abuse within the past five years or using drugs 3 months before the trial;
18. Subjects with underlying medical, psychiatric, psychological or other discomfort conditions, poor compliance, or who, as judged by the investigator, are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-27 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time zero to the time of the last quantifiable plasma concentration of the period (AUC0-last) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation) of AUC0-last within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Area under the curve from time zero to infinity (AUC0-inf) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of AUC0-inf within [0.8, 1.25] range will be used to determine the result of bioequivalence.

SECONDARY OUTCOMES:
Peak concentration at each treatment period (Cmax,tp) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of Cmax,tp within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Peak concentration of the first dosing (Cmax) | 1 month
  Individual pirfenidone and 5-carboxyl-pirfenidone plasma concentration-time profile for each treatment period will be established.
Time to reach peak concentration of the first dosing (Tmax) | 1 month
  Individual pirfenidone and 5-carboxyl-pirfenidone plasma concentration-time profile for each treatment period will be established.
Terminal half-life (T1/2) | 1 month
  Individual pirfenidone and 5-carboxyl-pirfenidone plasma concentration-time profile for each treatment period will be established.
Elimination rate constant (λz) | 1 month
  The PK parameters of each subject were calculated for statistical analysis
Apparent clearance（CL/F） | 1 month
  The PK parameters of each subject were calculated for statistical analysis
Apparent volume of distribution（Vd/F） | 1 month
  The PK parameters of each subject were calculated for statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Cao Yu, Doctor, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No